CLINICAL TRIAL: NCT07127731
Title: REACH BP: REmote Physical ACtivity Intervention for High Blood Pressure Postpartum
Brief Title: REmote Physical ACtivity Intervention for High Blood Pressure Postpartum
Acronym: REACH BP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Principal Investigator, Natalie Cameron, Instructor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STU00224381; 25CDA1449707 (Other Grant/Funding Number: American Heart Association)
Record Dates: First submitted 2025-07-31; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Hypertension (HTN); Hypertension ,Pregnancy; Physical Activity
Keywords: hypertension; pregnancy; postpartum; physical activity
MeSH Terms: conditions — Hypertension; Hypertension, Pregnancy-Induced; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental)
  Interventions: Behavioral: Patient Portal Messaging; Behavioral: FitBit EHR Linkage
- Control Group (Active Comparator)
  Interventions: Behavioral: FitBit EHR Linkage

INTERVENTIONS:
Behavioral: Patient Portal Messaging — Participants will receive weekly messages via their patient portal including feedback on their step counts and step count goals based on data from their FitBits
  Arms: Experimental Group
Behavioral: FitBit EHR Linkage — Participants will receive FitBits and link this step count data with the Electronic Health Record (EHR)

SUMMARY:
The purpose of this intervention is to help new mothers who had elevated blood pressure during pregnancy become more physically active after birth. The investigators will connect data from FitBits to the electronic health record. Women will then get weekly messages with feedback and goals to help them stay active. The investigators will test if the intervention improves step counts and blood pressure after pregnancy. The investigators will also test if the intervention is feasible and enjoyed by postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* Delivery of a live birth at Northwestern Medicine 6-12 weeks prior
* Systolic blood pressure 120-139 or diastolic blood pressure 80-89 during the first 20 weeks of gestation
* Low self-reported physical activity levels
* Able to access the internet at least weekly
* Have patient portal account or willing to set one up
* Willing to wear a FitBit
* Spoken and written English or Spanish language fluency

Exclusion Criteria:

* Medical contraindications to participating in a structured physical activity program
* Currently participating in a structured physical activity or weight loss program
* Hypertensive disorder of pregnancy (e.g., preeclampsia, gestational hypertension, eclampsia)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2027-04 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Recruitment | From enrollment to the end of the 24 week intervention
  Number of participants enrolled in the intervention
Feasibility of Participant Retention | At study weeks 12 and 24
  Percent of enrolled participants who continue to participate in the intervention
Feasibility of FitBit+EHR linkage | From enrollment to the end of the 24 week intervention
  Percent of intervention days FitBit data are linked to the Electronic Health Record
Feasibility of Intervention Messaging | From enrollment to the end of the 24 week intervention
  Percent of weekly messages that are read by participants
Acceptability of the Intervention | Study week 24
  Participants will fill out a survey to assess the extent to which they were satisfied with individual intervention components including FitBit usage, portal messaging, blood pressure and weight assessments, surveys, intervention length and intervention delivery. Each component will be rated on a 5-point Likert Scale in which 1 represents very dissatisfied (lowest score) and 5 represents very satisfied (highest score).

OTHER OUTCOMES:
Systolic Blood Pressure | Study weeks 0, 12 and 24
  Systolic blood pressure (mmHg)
Diastolic Blood Pressure | Study weeks 0, 12 and 24
  Diastolic Blood Pressure (mmHg)
Step Counts | Study weeks 0, 12 and 24
  Daily Mean Step Count from FitBits
Self Reported Physical Activity | Study weeks 0, 12 and 24
  Self-reported Metabolic Equivalent of a Task (MET)*hours per week based on responses to the Pregnancy Physical Activity Questionnaire
Body weight | Study weeks 0, 12 and 24
  Body weight (kg)
Height | Baseline
  Height in inches
Sleep | Study weeks 0, 12 and 24
  Mean hours of sleep per night
Diet | Study weeks 0, 12 and 24
  Adherence to Mediterranean diet assessed by the Mediterranean Eating Pattern for Americans Tool
Depression | Study weeks 0, 12 and 24
  Score on the Edinburgh Postnatal Depression Scale. Minimum Score: 0 (Least Depressed), Maximum Score: 30 (Most Depressed)
Perceived Stress | Study weeks 0, 12 and 24
  Score on the Perceived Stress Scale. Minimum Score: 0 (Least Perceived Stress), Maximum Score: 40 (Most Perceived Stress)
Perceived Anxiety | Study weeks 0, 12 and 24
  Score on the Generalized Anxiety Disorder - 7 Scale. Minimum Score: 0 (Little Anxiety), Maximum Score: 21 (Severe Anxiety)
Physical Activity Related Knowledge - Minutes Per Week | Study weeks 0, 12 and 24
  Participants will be asked a multiple choice question with 5 possible options about how many minutes per week of exercise is recommended by the government. One option will be considered the correct answer.
Blood Pressure Related Knowledge | Study weeks 0, 12 and 24
  Participants will be asked to write a response to the following question: Above which blood pressure does the American Heart Association say someone has hypertension?
Health Care Visits | From enrollment through the end of the 24 week intervention
  Number and type of healthcare visits attended
Sleep | Study weeks 0, 12 and 24
  Score on the PROMIS (Patient-Reported Outcomes Measurement Information System) Sleep Disturbance Short Form. Minimum Score: 8 (low levels of sleep disturbance; Maximum Score: 40 (high levels of sleep disturbance)
Physical Activity Counseling | From enrollment through the end of the 24 week intervention
  Number of times participant reports receiving physical activity counseling from a healthcare provider
FitBit Counseling | From enrollment through the end of the 24 week intervention
  Number of times participant reports discussing their FitBit data with a healthcare provider

IPD SHARING:
Plan to Share IPD: Yes
Any factual data that is needed for independent verification of research results will be made freely and publicly available in a repository as soon as possible, and no later than the time of an associated publication or 3/31/2028, whichever comes first.